CLINICAL TRIAL: NCT03619889
Title: The Effectiveness of the Pressure Release Technique on Masticatory and Neck Muscle Trigger Points in Patients With Chronic Myofascial Temporomandibular Disorder
Brief Title: The Effectiveness of a Physiotherapy Technique in Patients With Chronic Myofascial Temporomandibular Disorder
Acronym: TrP-TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gema Serrano-Hernanz, Principal Investigator, Clinical Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Geseher
Record Dates: First submitted 2018-05-27; First posted 2018-08-08 (Actual); Results first posted 2019-10-24 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Myofascial Pain Syndrome; Temporomandibular Disorder
Keywords: Chronic Pain; Physical Therapy modalities
MeSH Terms: conditions — Myofascial Pain Syndromes; Temporomandibular Joint Disorders; Chronic Pain | interventions — Myofascial Release Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: clinical trial, prospective, randomized and experimental with masking of the statistician and the participants
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants don´t know to which group are assigned The statistical assessor don´t know the aim of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham simulation group (Sham Comparator): A simulation of the pressure release technique, applying a soft pressure or contact in the same muscles sites or trigger points than in the intervention group.
  Interventions: Other: Sham
- Pressure release technique group (Experimental): The release pressure technique is applied in the trigger points of masticatory and neck muscles (upper trapezius, sternal and clavicular sternocleidomastoid, deep and superficial masseter, posterior, medium and anterior temporalis.
  Interventions: Other: Manual pressure release technique on trigger points.

INTERVENTIONS:
Other: Manual pressure release technique on trigger points. — A specific pressure is applied on trigger points of masticatory and neck muscles between pain pressure threshold and pain tolerance (7-8 visual analog scale).
  Other Names: Myofascial release
  Arms: Pressure release technique group
Other: Sham — A simulated pressure release technique is applied around masticatory and neck muscles.
  Other Names: Placebo
  Arms: Sham simulation group

SUMMARY:
Participants with chronic orofacial pain caused by masticatory and neck muscles will be distributed in two groups, both followed with the same occlusal and self-care treatment. The experimental group will receive 5 sessions of physiotherapy applying a specific pressure on the trigger points while the control group will receive placebo through a simulation of the same technique. Orofacial perceived pain, pain pressure thresholds, catastrophizing, kinesiophobia, cervical disability, depression and anxiety will be evaluated at baseline, immediately after treatment and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years.
* Patients diagnosed of myofascial TMD with at least one TrP with referred pain.
* TMD patients with a current complaint of myofascial pain with more than 6 months of evolution.
* Patients with myofascial TMD initially treated with splint currently used, that has not been modified in the last 6 months, without improvement.

Exclusion Criteria:

* Patients treated with occlusal splint recently modified.
* Patients with acute TMJ diseases.
* Patients with systemic disease, neurological and muscular diseases.
* Patients with psychiatric or psychological disorders.
* Patients with cervical disc hernia and acute whiplash injury.
* Changes in the painkillers intake during the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gema Serrano-Hernanz, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Odontology Faculty. Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serrano-Hernanz G, Angulo-Carrere T, Ardizone-Garcia I, Svensson P, Alvarez-Mendez AM. Pressure release technique versus placebo applied to cervical and masticatory muscles in patients with chronic painful myofascial temporomandibular disorder: A randomised clinical trial. J Oral Rehabil. 2023 Sep;50(9):782-791. doi: 10.1111/joor.13490. Epub 2023 May 25. PMID 37163204

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Pressure Release Technique GROUP: The Pressure Release Technique is applied in the trigger points of masticatory and neck muscles (upper trapezius, sternal and clavicular sternocleidomastoid, deep and superficial masseter, posterior, medium and anterior temporalis.
  Manual pressure release technique on trigger points.: A specific pressure is applied on trigger points of masticatory and neck muscles between pain pressure threshold and pain tolerance (7-8 visual analog scale).
Period: Overall Study
Arm/Group | Sham Simulation GROUP | Manual Pressure Release Technique GROUP
Started | 37 | 37
Completed | 35 | 37
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: A simulation of the pressure release technique, applying a soft pressure or contact in the same muscles sites or trigger points than in the intervention group.
  Sham: A simulated pressure release technique is applied around masticatory and neck muscles.
- Intervention Group: The release pressure technique is applied in the trigger points of masticatory and neck muscles (upper trapezius, sternal and clavicular sternocleidomastoid, deep and superficial masseter, posterior, medium and anterior temporalis.
  Manual pressure release technique on trigger points.: A specific pressure is applied on trigger points of masticatory and neck muscles between pain pressure threshold and pain tolerance (7-8 visual analog scale).
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 65
  >=65 years | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 37 | 72
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Changes of Perceived Pain Between Three Time Points (Baseline, Post-treatment, and 3 Months Later) and Between Groups (Sham Simulation and Pressure Release Technique)
Description: The Visual Analogue Scale (0-10) was used, 0 representing no pain/better outcome, and 10 representing unbearable pain/worst outcome.
  the clinical minimum relevance outcome is at least a change of 1.2 points in the scale.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | -1.03 (0.82) | -2.30 (1.16)
  value at 3 months later minus value at baseline | -0.77 (0.88) | -2.84 (1.94)
  value at 3 months later minus value at post-treatm | 0.26 (0.12) | -0.54 (0.31)
Statistical Analysis 1: Comparison: Pressure Release Technique GROUP; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Sham Simulation GROUP; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -1.2

2. Secondary Outcome: Changes of Pain Pressure Thresholds Anterior Temporalis
Description: An algometer Wagner Force One FDX 50 was used, measured in kgf/cm^2, with 0 representing the lowest pain pressure threshold/worst outcome and as higher pain pressure threshold/ as a better outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: kgf/cm^2
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
kgf/cm^2
  value at post-treatment minus value at baseline | -0.21 (0.36) | -0.48 (0.81)
  value at 3 months later minus value at baseline | -0.12 (0.24) | -0.40 (0.69)
  value at 3 months later minus value at post-treatm | 0.09 (0.38) | 0.08 (0.53)

3. Secondary Outcome: Changes in the Range of the Opening of the Mouth
Description: A calibrator Dentaurum München was used, measured in millimetres, with 0 representing no opening/worst outcome and as higher values/as a better outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
mm
  value at post-treatment minus value at baseline | -0.26 (5.81) | -4.27 (6.39)
  value at 3 months later minus value at baseline | -1.09 (6.59) | -5.22 (6.68)
  value at 3 months later minus value at post-treatm | -0.83 (1.81) | -0.95 (2.70)

4. Secondary Outcome: Changes in the Neck Disability
Description: The Neck Disability Index was used (0-50), with 0 representing no disability neck/best outcome and 50 maximum disability neck/worst outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 1.09 (2.67) | 5.78 (5.45)
  value at 3 months later minus value at baseline | 0.40 (1.61) | 5.40 (5.31)
  value at 3 months later minus value at post-treatm | -0.69 (2.48) | -0.38 (4.08)

5. Secondary Outcome: Changes in the Kinesiophobia
Description: The Tampa Scale for Kinesiophobia -11 was used (0-44), with 0 representing no kinesiophobia/best outcome and 44 representing the highest level of kinesiphobia/worst outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 1.80 (2.65) | 5.24 (4.49)
  value at 3 months later minus value at baseline | 1.83 (3.30) | 5.92 (4.94)
  value at 3 months later minus value at post-treatm | 0.03 (2.63) | 0.68 (2.43)

6. Secondary Outcome: Changes in the Catastrophizing
Description: The Pain Catastrophizing Scale was used (0-52), with 0 representing no catastrophizing/best outcome and 52 representing the highest level of catastrophizing/worst outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 2.14 (3.40) | 9.92 (7.68)
  value at 3 months later minus value at baseline | 0.80 (3.53) | 9.84 (7.50)
  value at 3 months later minus value at post-treatm | -1.34 (3.20) | -0.08 (4.67)

7. Secondary Outcome: Changes in the State Anxiety
Description: The State-Trait Anxiety Index was used, lower values represent a better outcome. State and Trait were evaluated individually, range of scores for each subtest is 20-80, with 20 representing no state anxiety/best outcome and 80 representing the highest level of state anxiety/worst outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 0.30 (0.93) | 1.59 (1.50)
  value at 3 months later minus value at baseline | 0.22 (0.82) | 1.53 (1.40)
  value at 3 months later minus value at post-treatm | -0.08 (0.55) | -0.05 (1.09)

8. Secondary Outcome: Changes in the State Depression
Description: The State-Trait Depression Inventory was used, lower values represent a better outcome. State and Trait were evaluated individually, range of scores for each subtest is 20-80, with 20 representing no state depression/best outcome and 80 representing the highest level of state depression/worst outcome
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 0.25 (0.68) | 0.74 (0.74)
  value at 3 months later minus value at baseline | 0.10 (0.60) | 0.75 (0.85)
  value at 3 months later minus value at post-treatm | -0.15 (0.43) | 0.01 (0.50)
Statistical Analysis 1: Comparison: Pressure Release Technique GROUP; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Sham Simulation GROUP vs Pressure Release Technique GROUP; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -0.65

9. Secondary Outcome: Changes in the Trait Anxiety
Description: The State-Trait Anxiety Index was used, lower values represent a better outcome. State and Trait were evaluated individually, range of scores for each subtest is 20-80, with 20 representing no trait anxiety/best outcome and 80 representing the highest level of trait anxiety/worst outcome.
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | -0.02 (0.34) | 0.68 (1.36)
  value at 3 months later minus value at baseline | -0.22 (0.67) | 0.59 (1.26)
  value at 3 months later minus value at post-treatm | -0.20 (0.73) | -0.09 (0.79)

10. Secondary Outcome: Changes in the Trait Depression
Description: The State-Trait Depression Inventory was used, lower values represent a better outcome. State and Trait were evaluated individually, range of scores for each subtest is 20-80, with 20 representing no Trait Depression/best outcome and 80 representing the highest level of Trait Depression/worst outcome
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
units on a scale
  value at post-treatment minus value at baseline | 0.15 (0.40) | 0.30 (0.60)
  value at 3 months later minus value at baseline | 0.07 (0.25) | 0.36 (0.61)
  value at 3 months later minus value at post-treatm | -0.07 (0.30) | 0.06 (0.76)

11. Secondary Outcome: Changes of Pain Pressure Thresholds Upper Trapezius
Description: as for outcome 2
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: kgf/cm^2
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
kgf/cm^2
  value at post-treatment minus value at baseline | -0.21 (0.36) | -0.48 (0.81)
  value at 3 months later minus value at baseline | -0.12 (0.24) | -0.40 (0.69)
  value at 3 months later minus value at post-treatm | 0.09 (0.38) | 0.08 (0.53)

12. Secondary Outcome: Changes of Pain Pressure Thresholds Sternal Sternocleidomastoid
Description: as for outcome 2
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: kgf/cm^2
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
kgf/cm^2
  value at post-treatment minus value at baseline | -0.14 (0.33) | -0.22 (0.48)
  value at 3 months later minus value at baseline | -0.08 (0.21) | -0.33 (0.70)
  value at 3 months later minus value at post-treatm | 0.06 (0.26) | -0.11 (0.64)

13. Secondary Outcome: Changes of Pain Pressure Thresholds Superficial Masseter
Description: as for outcome 2
Time Frame: Change from baseline in the scale at post-treatment and at 3 months later
Measure: Mean (Standard Deviation); unit: kgf/cm^2
Arm/Group | Sham Simulation GROUP | Pressure Release Technique GROUP
Number analyzed (Participants) | 35 | 37
kgf/cm^2
  value at post-treatment minus value at baseline | -0.23 (0.37) | -0.28 (0.66)
  value at 3 months later minus value at baseline | -0.21 (0.44) | -0.36 (0.59)
  value at 3 months later minus value at post-treatm | 0.02 (0.22) | -0.09 (0.54)

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed
Description: adverse events were not monitored/assessed
Groups:
- Sham Simulation GROUP: simulation of the pressure release technique
- Pressure Pain Technique GROUP: pressure release technique consists in aply pressure on muscular trigger points during 90 sec until the tissue barrier releases
Arm/Group | Sham Simulation GROUP | Pressure Pain Technique GROUP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03619889/Prot_SAP_ICF_000.pdf